CLINICAL TRIAL: NCT04391205
Title: Safety and Efficiency oh the Use of Midline Peripheral Venous Catheter (MIDES)
Brief Title: A Study to Investigate the Possible Causes of Secondary Effects During Use of Peripheral Midline Type Catheter in Patients Hospitalized in Different Care Settings
Acronym: MIDES
Status: Completed | Type: Observational
Sponsor: A.O.U. Città della Salute e della Scienza (Other)
Responsible Party: Principal Investigator, Dott.ssa RENATA MARINELLO, Principal Investigator, A.O.U. Città della Salute e della Scienza
Other Study IDs: 0041902
Record Dates: First submitted 2019-05-17; First posted 2020-05-18 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Upper Extremity Deep Vein Thrombosis, Secondary
Keywords: Midline; peripheral venous catheter; vascular access device; deep venous thrombosis
MeSH Terms: conditions — Upper Extremity Deep Vein Thrombosis; Venous Thrombosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Although the use of peripheral venous catheters (CVP) with brachial insertion with echo-guide (Midline) has increased significantly over the last 5-10 years, there are no sensitive data concerning complications in the literature during their use, particularly as regards incidence of thrombotic complication.The prospective observational study will enroll all the patients admitted to Home Health Hospitalization service, Geriatric Department and Intermediate Care service, to whom a Midline-type CVP will be placed for infusional therapy and who will give their consent to participate.

ELIGIBILITY:
Inclusion Criteria:

* Subjects admitted to wards adhering to the study (Home Health Hospitalization service, Geriatric Department and Intermediate Care service)
* Subjects submitted to Midline type venous catheter insertion

Exclusion Criteria:

* History of deep venous thrombosis or pulmonary embolism
* Be hospitalized for less than a week

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients were recruited in 3 different settings in the Molinette Hospital (Turin) - Home Health Hospitalization service, Geriatric Department and Intermediate Care service.
Sampling Method: Non-Probability Sample
Enrollment: 211 (Actual)
Dates: Start 2017-04-26 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Number of participants with Peripheral deep venous thrombosis (DVP) suspected with Compression ultrasound (CUS) and confirmed by echodoppler | Once a week from the implant day until CVP removal or patient discharge, whichever came first, assessed up to 40 days
  Deep vein thrombosis is investigated with Compression ultrasound (CUS) technique, scheduled once a week from the implant day or performed at the time of occurrence of device malfunctions or at the onset of symptoms resulting from thrombotic complications; echodoppler tecnique is used to confirm diagnosis of thrombosis.

CONTACTS AND LOCATIONS:
Overall Officials: Renata Marinello, MD, PhD, Principal Investigator — OAU Città della Salute e della Scienza di Torino, Turin, Italy
Locations (1):
- Marinello Renata, Turin, Italy